CLINICAL TRIAL: NCT00223678
Title: Mycophenolate Mofetil and Rapamycin as Secondary Intervention vs. Continuation of Calcineurin Inhibitors in Patients at Risk for Chronic Renal Allograft Failure
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Vanderbilt University Medical Center (Other)
Responsible Party: Principal Investigator, Anthony Langone, Anthony Langone M.D., Vanderbilt University Medical Center
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 000294
Record Dates: First submitted 2005-09-19; First posted 2005-09-22 (Estimated); Results first posted 2017-04-06 (Actual); Last update posted 2017-06-21 (Actual); Status verified 2017-05

CONDITIONS: Kidney Transplant
MeSH Terms: interventions — Sirolimus

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Active Comparator): pt will switch from calcineurin inhibitor (CYA, prograf) to Rapamycin
  Interventions: Drug: Rapamycin
- 2 (No Intervention): Patient will remain on calcineruin inhibitor

INTERVENTIONS:
Drug: Rapamycin — Rapamycin will start within 24 hours of last calcineurin inhibitors (Cya, Prograf). Initial dose of Rapamune 10mg will be given for 3 days and then dose will be adjusted to attain a target whole blood trough of 5-15
  Other Names: Sirolimus
  Arms: 1

SUMMARY:
A study to determine the effect on renal function in renal transplant patients with biopsy proven Chronic allograft nephropathy (CAN) nephropathy who are switched from a Calcinerin inhibitor (CI) triple drug regimen to a Rapamycin based triple drug regimen or maintained on their CI protocol

ELIGIBILITY:
Inclusion Criteria:

1. Patient is the recipient of a cadaveric or living donor renal transplant.
2. Patient was > 12 years of age at the time of transplant.
3. Patient is at least 3 months post-transplant.
4. Patient has been on a calcineurin inhibitor based immunosuppression since the transplant.
5. Patient has one of the following risk factors for chronic renal allograft failure:

   I. Serum creatinine > 2.0 mg/dL 3 months or later post-transplant in males patients.

   II. Serum creatinine > 1.7 mg/dL 3 months or later post-transplant in female patients.

   III. Serum > 30% increased over post discharge nadir.
6. Patients had a renal biopsy that shows chronic allograft nephropathy.
7. Patient or legal guardian had signed and dated an Institutional Review Board (IRB) approved informed consent document and is willing and able to follow study procedures.
8. If female and of child bearing potential, patient has a negative pregnancy test and agrees to practice effective birth control while receiving mycophenolate mofetil (MMF), Rapamycin and other immunosuppressants.

   -

Exclusion Criteria:

1. Patient is the recipient of a solid organ transplant other than the kidney.
2. Patient is dialysis dependent.
3. Patient has recurrence of primary renal disease, or de novo renal disease.
4. Patient has an estimated creatinine clearance <25ml/min calculated using the Cockcroft/Gault formula.
5. Patient has changed maintenance immunosuppressant therapy (e.g., azathioprine to MMF) within three months of randomization.
6. Baseline biopsy shows acute rejection Banff Grade > Class 2 (IIB).
7. Patient required anti-lymphocyte therapy to treat rejection found on baseline biopsy.
8. Patient has received an investigational immunosuppressant within three months.
9. Patient is pregnant or lactating.
10. Patient is a known carrier of any of the HIV viruses.
11. Patient has known hypersensitivity to Rapamycin, or any of the excipients of the drug.

Min Age: 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2000-06; Primary Completion 2009-10 (Actual); Study Completion 2009-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Anthony Langone, M.D., Principal Investigator — Vanderbilt University
Locations (1):
- Vanderbilt University, Nashville, Tennessee, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- Rapamycin: pt will switch from calcineurin inhibitor (CYA, prograf) to Rapamycin
  Rapamycin: Rapamycin will start within 24 hours of last calcineurin inhibitors (Cya, Prograf). Initial dose of Rapamune 10mg will be given for 3 days and then dose will be adjusted to attain a target whole blood trough of 5-15
- CYA/Prograf: Patient will remain on calcineurin inhibitor,CYA/Prograf
Period: Overall Study
Arm/Group | Rapamycin | CYA/Prograf
Started | 13 | 7
Completed | 13 | 7
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Population: approximately 30 patients will be randomized in a 2:1 ratio: two patients will be converted to Rapamycin-based immunosuppression for each patient randomized to continue calcineurin inhibitor based immunosuppression.
Groups:
- Total: Total of all reporting groups
Arm/Group | Rapamycin | CYA/Prograf | Total
Number analyzed (Participants) | 13 | 7 | 20
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 13 | 7 | 20
  >=65 years | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5 | 1 | 6
  Male | 8 | 6 | 14
Region of Enrollment [Number; unit: participants]
  United States | 13 | 7 | 20

OUTCOME MEASURES:

1. Primary Outcome: Graft Survival
Time Frame: 3 years
Measure: Median (95% Confidence Interval); unit: participants
Groups:
- Rapamycin Group: pt will switch from calcineurin inhibitor (CYA, prograf) to Rapamycin.Rapamycin: Rapamycin will start within 24 hours of last calcineurin inhibitors (Cya, Prograf). Initial dose of Rapamune 10mg will be given for 3 days and then dose will be adjusted to attain a target whole blood trough of 5-15
- CNI Group: Patient will remain on calcineurin inhibitor with a low target serum levels 50ng/ml to 125ng/mg 12 hour trough
Arm/Group | Rapamycin Group | CNI Group
Number analyzed (Participants) | 13 | 7
participants | 13 [1 to 36] | 7 [1 to 36]
Statistical Analysis 1: Comparison: Rapamycin Group vs CNI Group; Test type: Superiority or Other; p = 0.849, Log Rank

ADVERSE EVENTS:
Arm/Group | Rapamycin Group | CNI Group
Serious Adverse Events (participants affected / at risk) | 9/13 | 2/7
Other Adverse Events (participants affected / at risk) | 0/13 | 0/7
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Rapamycin Group (N=13) | CNI Group (N=7)
pneumonia (Respiratory, thoracic and mediastinal disorders) | 4 (4) | 1 (1)
acute kidney failure (Renal and urinary disorders) | 2 (2) | 1 (1)
dehydration (Vascular disorders) | 1 (1) | 0 (0)
hip replacement (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
acute rejection (Renal and urinary disorders) | 1 (1) | 0 (0)
total abdominal hysterectomy and salpingectomy (Reproductive system and breast disorders) | 1 (1) | 0 (0)
anemia (Blood and lymphatic system disorders) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less